CLINICAL TRIAL: NCT03800017
Title: Investigating the Role of Skeletal Muscle Dysfunction on Dyspnea and Exercise Intolerance in Interstitial Lung Disease
Brief Title: Skeletal Muscle Function in Interstitial Lung Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Jordan Guenette, Associate Professor, University of British Columbia
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: H18-02059
Record Dates: First submitted 2018-11-21; First posted 2019-01-10 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Interstitial Lung Disease; Idiopathic Pulmonary Fibrosis; Hypersensitivity Pneumonitis; Scleroderma; Nonspecific Interstitial Pneumonia
MeSH Terms: conditions — Lung Diseases, Interstitial; Idiopathic Pulmonary Fibrosis; Alveolitis, Extrinsic Allergic; Scleroderma, Diffuse

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyperoxia (Experimental): During exercise on visit 4, participants in both groups (i.e., ILD patients and controls) will breathe supplemental oxygen (i.e., 60% oxygen) during constant-load exercise.
  Interventions: Biological: Hyperoxia
- Healthy Controls (Placebo Comparator): During exercise on visit 3, participants in both groups (i.e., ILD patients and controls) will breathe ambient air (i.e., 20.93% oxygen) during constant-load exercise.
  Interventions: Biological: Hyperoxia

INTERVENTIONS:
Biological: Hyperoxia — Participants breathe 60% oxygen during exercise

SUMMARY:
Dyspnea (i.e. breathlessness) and exercise intolerance are common symptoms for patients with interstitial lung disease (ILD), yet it is not known why. It has been suggested that muscle dysfunction may contribute to dyspnea and exercise intolerance in ILD. Our study aims to: i) examine differences in the structure and function of the leg muscles in ILD patients, ii) determine if leg muscle fatigue contributes to dyspnea and exercise limitation in patients with ILD, and iii) determine the effects of breathing extra oxygen on leg muscle fatigue, as well as ability to exercise in ILD patients.

DETAILED DESCRIPTION:
PURPOSE:

The primary purpose of the proposed work is to characterize skeletal muscle function in patients with interstitial lung disease (ILD), and to determine the physiological and sensory consequences of impaired skeletal muscle function in ILD during exercise.

HYPOTHESES:

The hypotheses are threefold; i) patients with ILD will have impaired skeletal muscle function when compared to healthy controls, ii) impairments in skeletal muscle function predispose ILD patients to exercise-induced quadriceps muscle fatigue, increase the perception of exertional dyspnea, as well as reduce exercise tolerance, and iii) delivery of supplemental oxygen during exercise mitigates exercise-induced quadriceps muscle fatigue, attenuates the perceived intensity of dyspnea, and improves exercise tolerance.

OBJECTIVE:

The objective of the proposed study is to comprehensively investigate skeletal muscle dysfunction in patients with ILD and characterize its impact on dyspnea and exercise tolerance. In doing so, the proposed work will be the first to comprehensively assess skeletal muscle function in patients with ILD as well as determine its functional consequences. The results will provide important insight into the putative role of skeletal muscle dysfunction on exercise limitation in patient with ILD.

JUSTIFICATION:

ILD refers to a diverse group of diseases that share common physiological characteristics resulting from inflammation and/or fibrosis of the lung parenchyma. ILD has an estimated prevalence of approximately 67-81 cases per 100 000 individuals. Given the heterogeneity of disease sub-types, it is difficult to determine a precise median survival for patients with ILD, however; in patients with idiopathic pulmonary fibrosis, the most common ILD sub-type, have a median survival of only 2-3 years from the time of diagnosis. For patients with ILD, dyspnea (i.e. breathlessness) is the most common symptom. Dyspnea can be extremely debilitating, particularly during physical exertion. The clinical significance of dyspnea in ILD is underscored by its strong correlation with quality of life and mortality. Patients attempt to minimize dyspnea by avoiding physical activity, resulting in deconditioning and an associated reduction in functional capacity. The importance of maintaining functional capacity is highlighted by the fact that ILD patients with the lowest physical activity levels have the lowest quality of life and the highest mortality. The effective management of dyspnea and exercise intolerance is therefore of critical importance when considering the management of patients with ILD.

The pathophysiological mechanisms of dyspnea and exercise intolerance in ILD are complex, multifactorial, and poorly understood. Indeed, relatively few studies that have adequately investigated the mechanistic basis of dyspnea and exercise intolerance in patients with ILD. It is generally agreed upon that exercise limitation in ILD is related to the combination of altered respiratory mechanics, gas exchange impairment, and circulatory limitation. However, it is assumed that dyspnea and exercise intolerance are exclusively related to the respiratory and circulatory impairment associated with the pathogenesis of ILD. While this assumption is reasonable, it ignores the potentially crucial role of skeletal muscle dysfunction as a source of dyspnea and exercise intolerance. Recent experimental evidence indicates that skeletal muscle dysfunction contributes to both dyspnea and exercise intolerance in COPD.

A growing body of literature supports the notion that skeletal muscle dysfunction is common in ILD. While the precise mechanisms remain unclear, several well-established skeletal muscle dysfunction-promoting factors are present in many ILD patients, including: chronic hypoxaemia, oxidative stress, pulmonary and systemic inflammation, physical deconditioning, malnutrition, and corticosteroid use. These factors may act individually or synergistically to impair skeletal muscle function by causing muscle atrophy, mitochondrial dysfunction, a reduction in type I muscle fibre proportion, and increases in intramuscular fat. To our knowledge, there is limited imaging data of skeletal muscle morphology in ILD, and assessments of skeletal muscle oxidative capacity, and contractile function have not been concurrently obtained. If present, skeletal muscle dysfunction likely reduces locomotor muscle oxidative capacity, leading to premature fatigue, increased dyspnea, and diminished exercise tolerance. Most importantly, there is no data on the physiological effects of skeletal muscle fatigue and dysfunction on dyspnea and exercise capacity nor whether targeted treatment options such as supplemental oxygen (O2) delivery can attenuate muscle fatigue.

Accordingly, the aims of the proposed research are threefold: i) to characterize skeletal muscle function in patients with ILD compared to healthy controls, ii) to determine the influence of skeletal muscle dysfunction on dyspnea, fatigue, and exercise intolerance in patients with ILD compared to healthy controls, and iii) to determine if improving exercise tolerance using supplemental oxygen relieves exercise-induce skeletal muscle fatigue in ILD patients.

RESEARCH DESIGN:

Experimental hypotheses tested using combination of research designs. To test the hypotheses i) and ii), the investigators will use a cross sectional design. To test hypothesis iii), the investigators will use a single-blind placebo-controlled study design.

METHODS Participants will report to the laboratory on four separate occasions separated by a minimum of 48 hours, and each visit will last ~2-3 hours.

Visit 1:

Participants will complete medical history screening, complete a series of questionnaires concerning chronic activity-related dyspnea, quality of life, and physical activity. Participants will then have their height and weight measured and perform pulmonary function testing. Finally, participants will perform a symptom limited incremental cycle exercise test. Detailed physiological and sensory measurements will be obtained immediately before and throughout the incremental cycle exercise test.

Visit 1 will be intended to characterize participant's pulmonary function and exercise capacity.

Visit 2:

Participants will undergo a magnetic resonance imaging scan to assess the volume and the fat percentage of their quadriceps muscles They will then perform a series of tests aimed at evaluating their quadriceps muscle function, including: i) assessment of maximum voluntary quadriceps muscles strength, and ii) the non-invasive assessment of the oxidative capacity of their quadriceps muscle using near-infrared spectroscopy.

Data from visit 2 will be used to address hypothesis 1 by characterizing participant's quadriceps muscle function.

Visits 3:

Participants will perform a constant-load exercise test to exhaustion while breathing ambient air (i.e., 20.93% oxygen). The work load will be set at 75% of the highest work rate achieved during the incremental exercise test performed during visit 1.

Data from visits 3 and 4 will be used to address hypothesis 2 by characterizing the effect of exercise on skeletal muscle fatigue in patients with ILD and healthy controls.

Visit 4:

Participants will perform a constant-load exercise test while breathing supplemental oxygen (i.e., 60% oxygen). The work load will be set at 75% of the highest work rate achieved during the incremental exercise test performed during visit 1 and the test will be terminated once participants reach the same time that they achieved during the constant-load exercise test on Day 3.

Data from visit 4 will be used to address hypothesis 3 by determining if supplemental oxygen can be used to alleviate exercise-induced skeletal muscle fatigue in patients with ILD and healthy controls.

ELIGIBILITY:
Inclusion Criteria for ILD Patients:

* Age 40-80 years (inclusive)
* A multidisciplinary diagnosis of idiopathic pulmonary fibrosis (IPF), idiopathic fibrotic nonspecific interstitial pneumonia (NSIP), chronic hypersensitivity pneumonitis (HP), or unclassifiable ILD with a differential diagnosis that consists of the above diagnoses
* Fibrosis on high resolution computed tomography (HRCT): honeycombing, reticulation, or traction bronchiectasis
* Appropriate candidate for pulmonary rehabilitation
* 6 minute walk distance 50m or more
* Oxygen saturation ≥ 92% by pulse oximetry at rest while breathing room air
* Clinically stable for the preceding 6 weeks
* Can fluently read and write in English

Inclusion Criteria for Healthy Controls:

* Age 40-80 (inclusive)
* Normal pulmonary function (80-120% predicted)
* No lung or cardiovascular disease
* Can fluently read and write in English

Exclusion Criteria for the ILD patients:

* Contraindication to exercise testing (e.g. significant cardiovascular, musculoskeletal, neurological disease)
* Other significant extra-pulmonary disease that, based on clinical assessment, could impair exercise capacity and/or oxygenation
* Forced vital capacity (FVC) less than 50% or Diffusion capacity for carbon monoxide (DLCO) less than 25%
* Concurrent or recent participation (less than 6 months) in a pulmonary rehabilitation program
* Use of prednisone greater than 10 mg/day for more than 2 weeks within 3 months of the first study visit
* Significant emphysema (less than 10% volume on HRCT or FEV1/FVC less than 0.70)

Exclusion Criteria for Healthy Controls:

* Currently smoking or previously smoked more than 10 pack-years
* Any medical conditions that prevents them for exercising safely
* Cardiac pacemaker or any metal or electronic inside the body

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-08-07 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in standardized dyspnea score during the constant load exercise test (visit 3) | Dyspnea will be measured once every minute during exercise on visit 3 (up to 7 weeks after baseline) until participants reach volitional exhaustion (assessed for up to 30 minutes)
  Dyspnea rating, measured using the Borg 0-10 category ratio scale, will be assessed every 1 minute during the constant-load exercise test on visit 3.
Change in standardized dyspnea score during the constant load exercise test (visit 4) | Dyspnea will be measured once every minute during exercise on visit 4 (up to 8 weeks after baseline) until participants reach volitional exhaustion (assessed for up to 30 minutes)
  Dyspnea rating, measured using the Borg 0-10 category ratio scale, will be assessed every 1 minute during the constant-load exercise test on visit 4.
Change in leg muscle strength measured following the constant load exercise test (visit 3) | Leg muscle strength will be measured before and after exercise (assessed for up to 40 minutes) on visit 3 (up to 8 weeks after baseline)
  Leg muscle strength will be measured before (at rest) and 3 min after the constant-load exercise test on visit 3 using the femoral magnetic stimulation technique.
Change in leg muscle strength measured following the constant load exercise test (visit 4) | Leg muscle strength will be measured before and after exercise (assessed for up to 40 minutes) on visit 4 (up to 8 weeks after baseline)
  Leg muscle strength will be measured before (at rest) and 3 min after the constant-load exercise test on visit 4 using the femoral magnetic stimulation technique.

SECONDARY OUTCOMES:
Quadriceps muscle oxidative capacity measured using near-infrared spectroscopy | On visit 2, approximately 3 weeks post-baseline (visit 1)
  Quadriceps muscle oxidative capacity will measured using near-infrared spectroscopy. Parameters will be measured over 5 minutes once on visit 2
Quadriceps muscle volume measured using magnetic resonance imaging | On visit 2, approximately 3 weeks post-baseline (visit 1)
  Quadriceps muscle volume will be measured using magnetic resonance imaging. Parameters will be measured over 15 minutes once on visit 2

CONTACTS AND LOCATIONS:
Overall Officials: Jordan A Guenette, PhD, Principal Investigator — University of British Columbia
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No